CLINICAL TRIAL: NCT06101030
Title: Comparing Post Operative Utilization of Incentive Spirometry With and Without Electronic Patient Reminder
Brief Title: Comparing Use of Incentive Spirometry With and Without Reminder
Status: Recruiting | Type: Observational
Sponsor: Tidal Medical Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: InSee 202301
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Post Operative
Keywords: Incentive spirometry; Post Operative; compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Signal On: Patient Signals ON
  Interventions: Device: Signal On
- Signal Off: Patient Signals Off

INTERVENTIONS:
Device: Signal On — InSee monitor patient signals are on.
  Groups: Signal On

SUMMARY:
This study is designed to determine if patients using an incentive spirometer with visual and auditory signals will increase their use of the incentive spirometer and prevent lung complications.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the frequency of patients' use of physician ordered incentive spirometry increases with visual and auditory electronic encouragement (signals) compared to the no signal cohort.

Secondarily this study will correlate short term outcomes of study patients to known short term outcome data from the study site and published data to determine if there is a relationship between frequency of use and positive or outcomes or complications, as cited by peer reviewed literature.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following Inclusion criteria to be eligible for participation in the study:

* Patient has undergone a qualifying surgical procedure.
* Patient is aged 18 years or over.
* Patient has incentive spirometry ordered or incentive spirometry must be part of the study site's standard of care which is implemented by hospital staff.
* Patient is able to comply with all study required incentive spirometry instructions.
* Patient is without severe hearing or impaired visual acuity deficiency such that they cannot hear or see the audible and visual signal for the InSee monitor.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria at baseline will be excluded from study participation:

  * Vulnerable Populations (Pregnant, minors, prisoners, those with significantly reduced mental acuity).
  * Patients where incentive spirometry is inappropriate (patients with Tractotomy, patients who are hemodynamically unstable, patients in reverse isolation due to infection).
  * Patients with a history of prior non-compliance or the presence or history of psychiatric condition (including drug or alcohol addiction), or cognitive issue which would in the opinion of the investigator, make it difficult for the patient to comply with the study procedures or follow the investigators instructions.
  * Any medical condition that, in the opinion of the investigator, would place the patient at increased risk if they participated.
  * Any Physician determination that the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post Operative Inpatients prescribed incentive spirometry.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-09-03 (Estimated); Study Completion 2025-09-07 (Estimated)

PRIMARY OUTCOMES:
Number of successful inspiratory breaths attempts per day. | through hospitalization an average of 5 days
  successful inspiratory breaths is defined as achieving the goal tidal volume
Total number of inspiratory breaths achieved per day. | throughout hospitalization an average of 5 days
  Inspiratory breaths while using the incentive spirometer

SECONDARY OUTCOMES:
Time to achieve goal tidal volume. | throughout hospitalization an average of 5 days
  Time in to achieve prescribed goal inspiratory tidal volume.
Post operative length of O2 use. | throughout hospitalization an average of 5 days
  Length of time from surgery until 02 is discontinued.
Change in 02 flow rate. | throughout hospitalization an average of 5 days
  Change in 02 flow rate delivered to the patient.
inpatient Pulmonary complication rates. | throughout hospitalization an average of 5 days
  Pulmonary complications during hospitalization
Hospital discharge on O2. | throughout hospitalization an average of 5 days
  If a study patient is discharged on 02.
Changes in Inspiratory volume. | throughout hospitalization an average of 5 days
  Changes (- or +) in the inspiratory volume a patient is able to achieve.
Change in Inspiratory volume. | throughout hospitalization an average of 5 days
  Postoperative change in inspiratory volume
Readmission for pulmonary complication | 30 days after discharge
  Readmission for pulmonary complication up to 30 days after hospital discharge

OTHER OUTCOMES:
Intubation due to a respiratory diagnosis | throughout hospitalization an average of 5 days
  Postoperative Intubation due to a respiratory diagnosis during hospitalization
Reintubation due to a respiratory diagnosis | throughout hospitalization an average of 5 days
  Reintubation due to a respiratory diagnosis during hospitalization
ICU length of stay | throughout hospitalization an average of 5 days
  Postoperative length of stay in ICU
Inpatient hospital length of stay | throughout hospitalization an average of 5 days
  Postoperative length of stay in hospital
Change in SP02 | throughout hospitalization an average of 5 days
  Postoperative Change in SP02

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Study Director, M.D., Study Director — Tidal Medical Technologies
Locations (3):
- United States (3):
  - Tidal Reseach Site, Silver Spring, Maryland
  - Tidal Study Site, Rochester, Minnesota
  - Tidal Study Site, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eltorai AEM, Baird GL, Eltorai AS, Pangborn J, Antoci V Jr, Cullen HA, Paquette K, Connors K, Barbaria J, Smeals KJ, Agarwal S, Healey TT, Ventetuolo CE, Sellke FW, Daniels AH. Incentive Spirometry Adherence: A National Survey of Provider Perspectives. Respir Care. 2018 May;63(5):532-537. doi: 10.4187/respcare.05882. Epub 2018 Jan 23. PMID 29362219
- [Background] Sweity EM, Alkaissi AA, Othman W, Salahat A. Preoperative incentive spirometry for preventing postoperative pulmonary complications in patients undergoing coronary artery bypass graft surgery: a prospective, randomized controlled trial. J Cardiothorac Surg. 2021 Aug 24;16(1):241. doi: 10.1186/s13019-021-01628-2. PMID 34429138
- [Background] Alwekhyan SA, Alshraideh JA, Yousef KM, Hayajneh F. Nurse-guided incentive spirometry use and postoperative pulmonary complications among cardiac surgery patients: A randomized controlled trial. Int J Nurs Pract. 2022 Apr;28(2):e13023. doi: 10.1111/ijn.13023. Epub 2021 Oct 22. PMID 34676618